CLINICAL TRIAL: NCT00116142
Title: Docetaxel Plus 6-month Androgen Suppression and Radiation Therapy Versus 6-month Androgen Suppression and Radiation Therapy for Patients With High Risk Localized or Locally Advanced Prostate Cancer: A Randomized Controlled Trial
Brief Title: Hormone Suppression and Radiation Therapy for 6 Months With/Without Docetaxel for High Risk Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Anthony V. D'Amico, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-043
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Hormone Refractory; Metastatic; Localized; Locally Advanced; Prostate Cancer - High Risk Localized or Locally Advanced
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1: Androgen Suppression Therapy + Radiation Therapy (Other): Androgen Suppression Therapy and Radiation therapy
  Interventions: Drug: Androgen Hormonal Suppression and Radiation; Drug: Androgen Suppression Therapy and Radiation Therapy
- Arm 2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy (Experimental): Docetaxel plus androgen suppression therapy and radiation therapy
  Interventions: Drug: Docetaxel; Drug: Androgen Hormonal Suppression and Radiation; Drug: Androgen Suppression Therapy and Radiation Therapy

INTERVENTIONS:
Drug: Docetaxel — 60 mg/m² q 3 weeks for 3 cycle at the start of treatment followed by weekly Docetaxel at 20 mg/m² per week beginning at week one of radiation therapy and continuing for seven weeks.
  Other Names: Taxotere
  Arms: Arm 2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Drug: Androgen Hormonal Suppression and Radiation — Total Androgen Ablation and external beam radiation therapy
Drug: Androgen Suppression Therapy and Radiation Therapy — Total Androgen Ablation and External Beam Radiation Therapy

SUMMARY:
This randomized study is looking at the benefits of using docetaxel (chemotherapy) added to one of the standard treatments (radiation and hormones) for men with high-risk prostate cancer.

DETAILED DESCRIPTION:
Radiation therapy plus six months of hormone therapy is one standard way of treating men with high-risk prostate cancer. In this study, we want to see whether or not adding the chemotherapy drug docetaxel (Taxotere)will make this treatment more effective. Docetaxel has shown a benefit in median survival when given to men who have become resistant to hormonal therapy and in men who have metastatic prostate cancer (spread to other areas of the body).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer
* Clinical Tumor Category T1b, T1c, T2a and PSA greater than (>) 10 or Gleason score equal or greater than 4+3=7 or PSA velocity > 2.0 ng/ml per year and also eligible patients with tumor category T2c, T3a, T3b, or T4 as per 2002 AJCC guidelines. Any minor tertiary grade of Gleason 5; Biopsy Proven or Radiographic (erMRI Seminal Vesicle Invasion); Gleason = or > 3+4=7 with 50% or more cores positive
* Negative bone scan
* Lymph node assessment by CT or MR
* Adequate hematologic function (Blood Counts)
* Adequate liver functions (blood tests)
* ECOG performance Status 0 or 1
* Peripheral neuropathy must be =< grade 1
* PSA obtained within 3 months of entry

Exclusion Criteria:

* Prior history of malignancy that are < 5 years except for cancers found to be "in-situ" and would not likely impact a patient's life expectancy with appropriate medical management.
* Prior pelvic radiation therapy
* Prior hormonal therapy (up to 4 weeks prior to enrollment allowed)
* Individuals unable to tolerate lying still 5 - 10 minutes
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 90.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2005-06; Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V. D'Amico, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute and (Sanofi-Aventis Consortium), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayan M, Chen MH, Loffredo M, McMahon E, Moningi S, Orio PF, Nguyen PL, D'Amico AV. Elective Pelvic Lymph Node Radiation Therapy and the Risk of Death in Patients With Unfavorable-Risk Prostate Cancer: A Postrandomization Analysis. J Clin Oncol. 2024 Jul 20;42(21):2558-2564. doi: 10.1200/JCO.23.02394. Epub 2024 May 1. PMID 38691823
- [Derived] Sayan M, Huang J, Xie W, Chen MH, Loffredo M, McMahon E, Orio P, Nguyen P, D'Amico AV. Risk of Short-Term Prostate-Specific Antigen Recurrence and Failure in Patients With Prostate Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2336390. doi: 10.1001/jamanetworkopen.2023.36390. PMID 37801315
- [Derived] D'Amico AV, Xie W, McMahon E, Loffredo M, Medeiros S, Joseph D, Denham J, Kumar P, Bubley G, Sullivan M, Hellwig R, Carlos Vera J, Freter R, Jeffrey Baker W, Wong JY, Renshaw AA, Kantoff PW. Radiation and Androgen Deprivation Therapy With or Without Docetaxel in the Management of Nonmetastatic Unfavorable-Risk Prostate Cancer: A Prospective Randomized Trial. J Clin Oncol. 2021 Sep 10;39(26):2938-2947. doi: 10.1200/JCO.21.00596. Epub 2021 Jul 1. PMID 34197181
- [Derived] Guttilla A, Bortolus R, Giannarini G, Ghadjar P, Zattoni F, Gnech M, Palumbo V, Valent F, Garbeglio A, Zattoni F. Multimodal treatment for high-risk prostate cancer with high-dose intensity-modulated radiation therapy preceded or not by radical prostatectomy, concurrent intensified-dose docetaxel and long-term androgen deprivation therapy: results of a prospective phase II trial. Radiat Oncol. 2014 Jan 14;9:24. doi: 10.1186/1748-717X-9-24. PMID 24423462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9/21/2005 to 1/13/2015
Groups:
- Arm1: Androgen Suppression Therapy + Radiation Therapy: Androgen Suppression Therapy + Radiation therapy
  Weeks 1-9: total androgen suppression Weeks 10-17: total androgen suppression and external beam radiation Weeks 18-26: total androgen suppression
- Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
  Weeks 1-9: total androgen suppression and docetaxel 60 mg/m2/q3 weeks x 3 cycles Weeks 10-17: total androgen suppression + external beam radiation therapy + docetaxel 20 mg/m2/week beginning at week 10 x 7 cycles Weeks 18-26: total androgen suppression
Period: Overall Study
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Started | 175 | 175
Treated | 174 | 171
Completed | 156 | 155
Not Completed | 19 | 20
Not completed — Adverse Event | 8 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Physician Decision | 3 | 1
Not completed — Delayed Radiation Therapy | 1 | 0
Not completed — Patient could not tolerate docetaxel | 0 | 2
Not completed — Patient stopped due to depression | 0 | 1
Not completed — Patient stopped due to bilateral ruptured tendons | 0 | 1
Not completed — Patient didn't start due to diagnosis of colon cancer | 0 | 1
Not completed — Patient didn't start due to low platelet counts | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 85] | 66 [43 to 86] | 66 [43 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 175 | 175 | 350
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 139 | 132 | 271
  Black or African American | 4 | 5 | 9
  Asian | 3 | 1 | 4
  Other | 29 | 37 | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110 | 102 | 212
  Australia | 62 | 69 | 131
  New Zealand | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: 10-Year Restricted Mean Survival Time for Overall Survival
Description: Overall survival (OS) was measured from the date of random assignment to death from any cause, censored at the date of last follow-up in surviving patients. The 10-Year Restricted Mean Survival Time was calculated as the area under the Kaplan Meier plot for OS, from randomization to 10-years follow-up
Time Frame: Following the end of RT patients were seen for follow up every 6 months for 5 years and annually thereafter, 10 years.
Measure: Mean (Standard Error); unit: years
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Number analyzed (Participants) | 175 | 175
years | 8.82 (0.19) | 9.11 (0.15)

2. Secondary Outcome: 10-year Biochemical Recurrence (PSA Failure)
Description: Time to biochemical recurrence was defined as the time from date of random assignment to the earliest of PSA failure or initiation of salvage therapy, or censored at the date of last disease assessment for those without PSA failure. PSA failure was defined according to the 2006 RTOG-ASTRO Phoenix definition (i.e., A PSA rise by 2 ng/mL or more above the nadir).
  10-year biochemical recurrence rate was estimated from a competing risk model where non-prostate cancer death was counted as competing risk.
Time Frame: PSA was measured following the end of RT, then every 6 months for 5 years and annually thereafter, 10 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Arm1: Androgen Suppression Therapy + Radiation Therapy: Androgen Suppression Therapy and Radiation Therapy
  Weeks 1-9: total androgen suppression Weeks 10-17: total androgen suppression and external beam radiation Weeks 18-26: total androgen suppression
- Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy: Docetaxel + Androgen Suppression Therapy and Radiation Therapy
  Weeks 1-9: total androgen suppression and docetaxel 60 mg/m2/q3 weeks x 3 cycles
  Weeks 10-17: total androgen suppression + external beam radiation therapy + docetaxel 20 mg/m2/week beginning at week 10 x 7 cycles
  Weeks 18-26: total androgen suppression
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Number analyzed (Participants) | 175 | 175
percentage of subjects | 48 [39 to 55] | 54 [46 to 62]

3. Secondary Outcome: 10-year Prostate Cancer Mortality
Description: Measured from the date of random assignment to date of death from prostate cancer, or censored at the date of last follow-up in surviving patients. Patients who died due to other reasons were counted as competing risk in a competing risk model.
Time Frame: Following the end of RT patients were seen for follow up every 6 months for 5 years and annually thereafter, 10 years.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Number analyzed (Participants) | 175 | 175
percentage of subjects | 11 [7 to 17] | 15 [10 to 22]

4. Secondary Outcome: Number of Participants With Acute Adverse Events
Description: Adverse acute events were reported via the clinical database only for toxicities considered reportable via the SAE mechanism (those of grade 2 and grade 3 events that are unexpected and possibly, probably, or definitely related/associated with treatment; or all grade 4 and grade 5 events). Common Toxicity Criteria Volume 3.0 (CTCAE) is used for this study.
Time Frame: During study treatment or within 30 days of the last dose of study, up to 7.2 months from randomization
Population: Adverse acute events were evaluated in patients who received at least one dose of protocol treatment (174 out of 175 subjects in Arm1, 171 out of 175 subjects in Arm2).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Number analyzed (Participants) | 174 | 171
Participants | 18 | 46

5. Secondary Outcome: Number of Participants With Late Adverse Events, Any Grade and Attribution
Description: Late adverse events will be focused on GU/GI including Urinary/Fecal Incontinence, Hematuria, Diarrhea, Rectal Bleeding and other.
Time Frame: Every 6 months post radiation therapy for 5 years (+/-90 days), then annually, up to 13.9 years from randomization
Population: Adverse late event was evaluated in patients who received at least one dose of protocol treatment (174 out of 175 subjects in Arm1, 171 out of 175 subjects in Arm2).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
Number analyzed (Participants) | 174 | 171
Participants | 128 | 140

ADVERSE EVENTS:
Time Frame: Up to 13.9 years from randomization.
Description: Adverse acute events were reported via trial database only for those deemed reportable via the SAE mechanism (grade 2/3 events that are unexpected and possibly, probably, or definitely related to treatment; or all grade 4/5 events). Adverse late events include GU/GI toxicities. Adverse event was analyzed in patients who received at least one dose of study therapy (Arm1:174 out of 175 subjects, Arm2:171 out of 175). Mortality was analyzed in all randomized subjects by the intent-to-treat rule.
Arm/Group | Arm1: Androgen Suppression Therapy + Radiation Therapy | Arm 2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 45/175 | 44/175
Serious Adverse Events (participants affected / at risk) | 63/174 | 87/171
Other Adverse Events (participants affected / at risk) | 128/174 | 142/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1: Androgen Suppression Therapy + Radiation Therapy (N=174) | Arm 2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy (N=171)
Weight loss (Investigations) | 1 | 0
Perforation, colon (Gastrointestinal disorders) | 0 | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
Ulcer, duodenum (Gastrointestinal disorders) | 0 | 1
Cardiac-ischemia (Cardiac disorders) | 1 | 1
Cystitis (Renal and urinary disorders) | 1 | 1
Hot flashes (Vascular disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 2 | 1
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
C5 tetraplegia (Injury, poisoning and procedural complications) | 0 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1
Fever w/o neutropenia (General disorders) | 0 | 1
Gynecomastia (Reproductive system and breast disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 0 | 1
Infection w/ gr 3-4 neut, blood (Infections and infestations) | 0 | 1
Infection w/ unk ANC lung (Infections and infestations) | 0 | 1
Leukocytes (Investigations) | 0 | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 0 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Infection-other (Infections and infestations) | 0 | 2
Proctitis (Gastrointestinal disorders) | 1 | 3
Urinary retention (Renal and urinary disorders) | 4 | 3
Cardiac-other (Cardiac disorders) | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Erectile impotence (Reproductive system and breast disorders) | 3 | 6
Incontinence, anal (Gastrointestinal disorders) | 7 | 6
Rectum, hemorrhage (Gastrointestinal disorders) | 9 | 7
Incontinence urinary (Renal and urinary disorders) | 11 | 8
Neutrophils (Investigations) | 0 | 8
GI-other (Gastrointestinal disorders) | 10 | 9
Bladder, hemorrhage (Renal and urinary disorders) | 0 | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 9 | 17
Urinary frequency/urgency (Renal and urinary disorders) | 10 | 18
Renal/GU-other (Renal and urinary disorders) | 17 | 27
Bladder spasms (Renal and urinary disorders) | 1 | 0
Constitutional, other (General disorders) | 1 | 0
Death - sudden death (General disorders) | 1 | 0
Distention/bloating, abdominal (Gastrointestinal disorders) | 1 | 0
Endocrine-other (Endocrine disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Bladder, hemorrhage (Renal and urinary disorders) | 10 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1: Androgen Suppression Therapy + Radiation Therapy (N=174) | Arm 2: Docetaxel + Androgen Suppression Therapy + Radiation Therapy (N=171)
ALT, SGPT (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Bladder spasms (Renal and urinary disorders) | 1 | 0
Bladder, hemorrhage (Renal and urinary disorders) | 23 | 31
Cardiac-other (Cardiac disorders) | 0 | 1
Chest/thoracic pain NOS (General disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 24 | 17
Constitutional, other (General disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 42 | 50
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Erectile impotence (Reproductive system and breast disorders) | 5 | 4
Fracture (Injury, poisoning and procedural complications) | 0 | 1
GI-other (Gastrointestinal disorders) | 31 | 34
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Incontinence urinary (Renal and urinary disorders) | 35 | 52
Incontinence, anal (Gastrointestinal disorders) | 21 | 32
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 2 | 2
Infection w/ unk ANC wound (Infections and infestations) | 1 | 0
Infection-other (Infections and infestations) | 1 | 0
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 19 | 25
Nausea (Gastrointestinal disorders) | 0 | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 49 | 41
Renal/GU-other (Renal and urinary disorders) | 70 | 84
Rigors/chills (General disorders) | 0 | 1
Stenosis (incl anastomotic) small bowel (Gastrointestinal disorders) | 0 | 1
Testicle, pain (Reproductive system and breast disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 49 | 50
Urinary retention (Renal and urinary disorders) | 2 | 6
Vasovagal episode (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2005-05-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT00116142/Prot_SAP_000.pdf